CLINICAL TRIAL: NCT05012878
Title: Cerebral Blood Flow Regulation and Cognitive Function in Adults With Cardiovascular Disease - Influence of Exercise Training and Intensity
Brief Title: Cardiac Rehab and Cerebral Blood Flow Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Bruce Johnson, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20-010808
Record Dates: First submitted 2021-07-19; First posted 2021-08-19 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Randomized control trial comparing two cardiac rehabilitation exercise groups: 1) high intensity interval training; and 2) moderate intensity continuous training. There will also be an observational control group who decline participation in cardiac rehabilitation, and an observational cardiac rehabilitation group who participate in cardiac rehabilitation but decline randomization. There is also a healthy control group without cardiovascular disease for baseline comparison only (no intervention).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Cardiac rehabilitation - High intensity interval training (HIIT) (Experimental): Patients attending cardiac rehabilitation randomized to HIIT.
  Interventions: Behavioral: Cardiac rehabilitation - high intensity interval training (HIIT)
- Cardiac rehabilitation - Moderate intensity continuous training (MICT) (Active Comparator): Patients attending cardiac rehabilitation randomized to MICT.
  Interventions: Behavioral: Cardiac rehabilitation - moderate intensity continuous training (MICT)
- Cardiac rehabilitation - control (Placebo Comparator): The control group (12 week period) will include participants who have declined cardiac rehabilitation.
  Interventions: Behavioral: Cardiac rehabilitation - control
- Healthy control group (No Intervention): Healthy age-matched adults without cardiovascular disease, who will complete baseline assessments only. No intervention period.
- Cardiac rehabilitation - observational (Other): This observational group will include patients who are completing an exercise-based cardiac rehabilitation program in line with standard care but are not part of the randomized exercise protocol groups (HIIT or MICT). Participants in this group will be combined with HIIT and MICT (as exercise-based cardiac rehabilitation group) for Aims 1b and 2b.
  Interventions: Behavioral: Cardiac rehabilitation - observational

INTERVENTIONS:
Behavioral: Cardiac rehabilitation - high intensity interval training (HIIT) — During cardiac rehabilitation (12-weeks, 3 sessions/week), exercise training will comprise of 4x4-min high intensity aerobic intervals at a rating of perceived exertion 15-17 (hard to very hard), interspersed by a 3-min active recovery at a rating of perceived exertion 11-13 (fairly light to somewhat hard). Warm-up (4-min) and cool-down (3-min) at a light intensity.
  Other Names: CR-HIIT
  Arms: Cardiac rehabilitation - High intensity interval training (HIIT)
Behavioral: Cardiac rehabilitation - moderate intensity continuous training (MICT) — During cardiac rehabilitation (12-weeks, 3 sessions/week), exercise training will comprise of 34-min of continuous aerobic exercise at a rating of perceived exertion 11-13 (fairly light to somewhat hard). Warm-up (3-min) and cool-down (3-min) at a light intensity.
  Other Names: CR-MICT
  Arms: Cardiac rehabilitation - Moderate intensity continuous training (MICT)
Behavioral: Cardiac rehabilitation - control — Participants will receive exercise advice in line with usual hospital discharge procedures. This involves exercise physiologists providing verbal and written information on achieving the national physical activity guidelines (150min/week of moderate intensity exercise) 60 and range of movement exercises for surgical patients with sternotomy. However, no structured or supervised exercise training program or other contact with participants will be provided after hospital discharge, to reflect the usual care process for patients that decline cardiac rehabilitation.
  Other Names: CR-Control
  Arms: Cardiac rehabilitation - control
Behavioral: Cardiac rehabilitation - observational — During cardiac rehabilitation (12-weeks), program frequency and exercise training protocol will align with clinical care decisions and/or patient choice rather than random assignment.
  Other Names: CR-Observational
  Arms: Cardiac rehabilitation - observational

SUMMARY:
This study is being done to better understand the influence of cardiovascular disease on brain blood flow regulation and cognitive function, determine whether exercise-based cardiac rehabilitation can lead to better regulation of brain blood flow that may help to improve or maintain cognitive function, and determine whether exercise intensity influences changes in brain blood flow regulation and cognitive function.

DETAILED DESCRIPTION:
This study will investigate the influence of exercise training and intensity (as part of cardiac rehabilitation) on improving cerebral blood flow regulation and cognitive function following a cardiac event. This will be a randomized control trial, recruiting adults in mid-life (years 40-65) with coronary artery disease, enrolling in cardiac rehabilitation following a cardiac-related hospital admission. Patients that enroll in the Mayo Clinic cardiac rehabilitation will be randomized 1:1 to high intensity interval training (HIIT) or moderate intensity continuous training (MICT), with stratification for sex and coronary artery bypass graft surgery. Patients that decline enrollment in cardiac rehabilitation will be recruited as an observational control group, which will be matched to the intervention groups by age decade, sex, BMI category, and surgical status. Patients that enroll in cardiac rehabilitation but decline randomization will be recruited as an observational cardiac rehabilitation group. A healthy control group without cardiovascular disease will also be recruited for baseline comparison of outcome measures.

ELIGIBILITY:
Inclusion Criteria for Patients with Cardiovascular Disease:

* Aged 40-years and older.
* Eligible for cardiac rehabilitation following a cardiac-related hospital admission, coronary artery disease (including angina, myocardial infarction, percutaneous coronary intervention, or coronary artery bypass graft surgery).

Inclusion Criteria for Healthy controls:

* Aged 40-years and older.
* Never been diagnosed with cardiovascular disease or coronary artery disease.
* No history of cardiovascular disease risk factors including hypertension, hyperlipidemia, diabetes, obesity (body mass index > 30) or smoking.
* Current body mass index < 30kg/m2

Exclusion Criteria for participants in randomized cardiac rehabilitation groups (HIIT & MICT) :

* Known cerebrovascular or neurological disease
* Known moderate-severe respiratory disease, pregnancy,
* Orthopedic limitations affecting exercise capability
* Unable to read and speak English
* Unable to complete study-related activities
* Contraindications to hypercapnia
* Contraindications to maximal exercise testing
* MRI incompatible devices
* Unwillingness to undergo MRI scan (e.g. due to anxiety or claustrophobia).

Exclusion Criteria for participants in the observational control group and observational cardiac rehabilitation group:

* Known cerebrovascular or neurological disease
* Known moderate-severe respiratory disease, pregnancy,
* Unable to read and speak English
* Unable to complete study-related activities
* Contraindications to hypercapnia
* MRI incompatible devices
* Unwillingness to undergo MRI scan (e.g. due to anxiety or claustrophobia)

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2025-04-23 (Actual)

PRIMARY OUTCOMES:
Cerebral blood flow regulation (as cerebrovascular reactivity) | Baseline and follow-up at 3-months
  Measured as the change in cerebral blood flow during a stepped protocol of increases in inhaled carbon dioxide concentrations. Reactivity will be measured as the regression slope of cerebral blood flow velocity (cm per second) per mmHg increase in end-tidal carbon dioxide.

SECONDARY OUTCOMES:
Cognitive function | Baseline and follow-up at 3-months
  The main domains of cognitive function assessed using a neuropsychometric testing battery will be executive function, processing speed, and memory. Scores from these domains will be combined as the NIH Toolbox Fluid composite score, and assessed for change from baseline to follow-up. Analyses will also be completed for each separate cognitive domain.

OTHER OUTCOMES:
Cerebral blood flow regulation (as neurovascular coupling) | Baseline and follow-up at 3-months
  Measured as the change in cerebral blood flow during a visual stimulus
Cerebral blood flow regulation (as autoregulation) | Baseline and follow-up at 3-months
  Measured as the change in cerebral blood flow from seated position to standing position.
Cerebral blood flow regulation to exercise | Baseline and follow-up at 3-months
  Measured as the regression slope of cerebral blood flow per increase in cardiac output (L) during a staged submaximal exercise test to 75% of maximal heart rate.
Cerebral ventricular and white matter hyperintensity volumes | Baseline and follow-up at 3-months
  Measured using MRPAGE and FLAIR MRI. Expressed as percentage of total intracranial volume
Resting cerebral blood flow with MRI | Baseline and follow-up at 3-months
  Measured using arterial spin labelling MRI. Global cerebral blood flow will be expressed as the average of gray matter perfusion across all atlas regions.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce D Johnson, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No